CLINICAL TRIAL: NCT01652768
Title: PRESENCE Project: An Early Palliative Care Intervention for Patients With Malignant Brain Tumors and Their Primary Caregivers
Brief Title: PRESENCE Project: An Early Palliative Care Intervention in Brain Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research Cancelled
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1310
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Malignant Brain Tumors
Keywords: Malignant Brain Tumors; Malignant Glioma; High-grade Gliomas; Oncology; Cancer; Patient Caregiver; Caregiver Stress, Anxiety, Depression; Palliative Care Intervention
MeSH Terms: conditions — Glioma; Neoplasms; Caregiver Burden; Anxiety Disorders; Depression | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Usual Care Group (Active Comparator): Usual care is defined as standard post-operative care on a surgical unit in University Hospitals Case Medical Center. Discharge planning will be provided by the assigned in-patient social worker. Referrals to the assigned outpatient social worker will be made as appropriate. Patients and caregivers will be seen in the ambulatory medical oncology setting about three to six weeks after surgery, depending on post-operative recovery time. The research assistant will administer the research questionnaires at week one post-surgery and 8-10 weeks post surgery.
  Interventions: Other: Research Questionnaires
- Arm B: PRESENCE Intervention (Experimental): The unique features of the PRESENCE Project (PP) Intervention are 1) the early palliative care intervention (immediately post-op) provided by the new palliative care brain tumor team (Social worker, advanced practice nurse (APN), medical oncology registered nurse); 2) an educational information session for patients and caregivers; and 3) frequent (every two week and as needed) telephone or clinic visits during the first ten weeks post operatively (Figure 1). In usual care, the patient and caregiver receive little supportive care until they begin cancer treatment. The intervention provides aggressive supportive care from the time of diagnosis.
  Interventions: Other: Research Questionnaires; Other: Palliative Care Team; Other: Educational Information Session for Patients and Caregivers; Other: Contact every 2 weeks; Other: Follow-up Surgical Visit Session; Other: Medical and/or Radiation Oncology Appointment Session

INTERVENTIONS:
Other: Research Questionnaires — Hospital Anxiety and Depression Scale Pearlin & Schooler Caregiver Mastery Caregiver Assessment Tool Patient/Caregiver Satisfaction Survey
Other: Palliative Care Team — Week 1: Early palliative care intervention (immediately post-op) provided by the new palliative care brain tumor team (Social worker, advanced practice nurse (APN), medical oncology registered nurse).
  1. Introduce the palliative care team concept.
  2. Provide contact information for the palliative care team given
  3. Administer Initial Patient and Caregiver Psychosocial Assessments (Appendix A)
  4. Offer community resources to patient and caregiver (Appendix B)
  5. Provide additional resources/referrals for any needs that are identified by patient or care partner during initial psychosocial assessment
  6. Provide supportive care
  Arms: Arm B: PRESENCE Intervention
Other: Educational Information Session for Patients and Caregivers — Provide an educational class "Moving Forward: Facing a Brain Tumor Diagnosis" for patient and caregiver Week 5 through 7: The PRESENCE Project Social Worker and oncology RN will provide an educational class.
  Intervention (Length of time for class = 2 hours):
  1. Provide an educational class "Moving Forward: Facing a Brain Tumor Diagnosis" for patient and caregiver.
  2. Provide additional resources/referrals for any needs that are identified by patient or care partner during the educational class.
  3. Provide supportive care.
  Arms: Arm B: PRESENCE Intervention
Other: Contact every 2 weeks — The PRESENCE Project APN and/or Presence Project Social Worker will contact the patient and caregiver via telephone or office visit every two weeks and as needed until the second medical oncology visit.
  (Anticipated length of time for phone intervention or visit is 20 minutes; however, length of time for intervention is tailored to the patient and caregiver's needs):
  1. Administer Patient and Caregiver Follow-up Assessment
  2. Provide pain and/or symptom management intervention for any issues identified during the follow-up assessment
  3. Provide resources/referrals for any needs identified during the social work follow-up assessment
  4. Provide supportive care
  Arms: Arm B: PRESENCE Intervention
Other: Follow-up Surgical Visit Session — The PRESENCE Project APN will meet with patient and caregiver at the surgical follow-up visit, approximately two weeks after surgery.
  Intervention (Anticipated length of time for visit is about 30 minutes; however length of time for intervention is tailored to the patient and caregiver's needs):
  1. Administer Patient and Caregiver Follow-up Assessment
  2. Administer Symptom Assessment Tool
  3. Provide pain and/or symptom management intervention
  4. Provide supportive care
  Arms: Arm B: PRESENCE Intervention
Other: Medical and/or Radiation Oncology Appointment Session — The PRESENCE Project APN and/or Presence Project Social Worker will meet with patient and caregiver at the first medical and/or radiation oncology appointment (weeks 3 and 4).
  Intervention (Anticipated length of time for visit is about 30 minutes; however length of time for intervention is tailored to the patient and caregiver's needs):
  1. Administer Patient and Caregiver Follow-up Assessment
  2. Re-assess pain and/or symptom management issues and /or intervention
  3. Provide resources/referrals for any needs identified during the social work follow-up assessment
  4. Provide supportive care.
  Arms: Arm B: PRESENCE Intervention

SUMMARY:
The purpose of this pilot study is to investigate the feasibility of an early palliative care intervention (PRESENCE: Providing Resources Education, Support, and Enabling New brain tumor patients to Cope Effectively) and the effect of the intervention on patient and caregiver distress.

DETAILED DESCRIPTION:
Patients and caregivers will be enrolled in two phases. Phase I is a qualitative study exploring the experience of primary caregivers of patients with a new diagnosis of malignant brain tumor during the first 10 weeks of the diagnosis and beginning treatment process. During Phase I, only caregivers patients with a malignant brain tumor who are at least two months and not more than six months into treatment at the Seidman Cancer Center (SCC)will be enrolled. They will be asked to participate in a qualitative interview to describe the newly diagnosed experience (diagnosis through first 10 weeks of treatment) of having a loved one with a malignant brain tumor.

A convenience sample of 20 patients and their primary caregivers will be enrolled for Phase II of this pilot project. The first ten patients and caregivers enrolled will receive usual care (Phase II, Arm A). Usual care is defined as standard post-operative care on a surgical unit in University Hospitals Case Medical Center. Discharge planning will be provided by the assigned in-patient social worker. Referrals to the assigned outpatient social worker will be made as appropriate. Patients and caregivers will be seen in the ambulatory medical oncology setting about three to six weeks after surgery, depending on post-operative recovery time.

The second ten patients and caregivers enrolled will receiving the intervention (Phase II, Arm B). The unique features of the PRESENCE Project (PP) Intervention are 1) the early palliative care intervention (immediately post-op) provided by the new palliative care brain tumor team (Social worker, advanced practice nurse (APN), medical oncology registered nurse); 2) an educational information session for patients and caregivers; and 3) frequent (every two week and as needed) telephone or clinic visits during the first ten weeks post operatively. In usual care, the patient and caregiver receive little supportive care until they begin cancer treatment. The intervention provides aggressive supportive care from the time of diagnosis.

RESEARCH OBJECTIVES:

1. To investigate the feasibility of an early palliative care intervention (PRESENCE: Providing Resources Education, Support, and Enabling New brain tumor patients to Cope Effectively) for patients newly diagnosed with a malignant brain tumor and their primary caregivers.
2. To explore the experience of being a caregiver of a patient newly diagnosed with a malignant brain tumor.
3. To determine the effect of the PRESENCE Intervention on patient and caregiver distress, anxiety, and depression.
4. To determine the effect of the PRESENCE Intervention on caregiver reaction (benefit and burden) and caregiver mastery.

ELIGIBILITY:
Inclusion Criteria for Caregivers (Phase I):

* are identified by the patient and/or caregiver as the "primary caregiver"
* were involved in caregiving during the first ten weeks following diagnosis at the SCC
* are capable of providing informed consent.

Exclusion Criteria for Caregivers (Phase I):

- include those whose are caring for patients who are in hospice or within 2 months of death, as this experience may influence their recollection of the diagnosis phase of the cancer trajectory.

Inclusion Criteria for Patients (Phase II):

* are newly diagnosed malignant brain tumor patients who are at University Hospitals and who are within a week of surgery
* are receiving on-going care at the Seidman Cancer Center
* are able to identify a primary caregiver involved in their care, support, and/or care planning
* are capable of providing informed consent.

Exclusion Criteria for Patients (Phase II):

- are those with a life expectancy of less than two months and/or those who are electing hospice care who will be receiving medical and or radiation oncology care outside of the Seidman Cancer Center.

Eligibility criteria for caregivers (Phase II)

* being identified by the patient as the "primary caregiver"
* capable of providing informed consent.
* Both the patient and caregiver must consent to be in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention will be measured by participant surveys. | 10 weeks
  Using the patient satisfaction tool, the researchers will report descriptive data on patient and caregiver satisfaction with the intervention and any burden associated with participating in the intervention. In addition, the ability to contact patients and caregivers on an every two week basis, patient and caregiver attendance at the educational program, and evaluations from the Moving Forward program will be tracked.

SECONDARY OUTCOMES:
Change in distress level | 10 weeks
  Using the patient satisfaction tool, the researchers will report descriptive data on patient and caregiver satisfaction with the intervention and any burden associated with participating in the intervention. In addition, the ability to contact patients and caregivers on an every two week basis, patient and caregiver attendance at the educational program, and evaluations from the Moving Forward program will be tracked.
Change in Anxiety level | 10 weeks
  Distress: Psychological distress is defined as "the general concept of maladaptive psychological functioning in the face of stressful life events" (Abeloff et al., 2000, p. 556). Distress is being measured as a global construct, using a distress thermometer as described by the National Comprehensive Cancer Network (NCCN) Guidelines (Holland & Alici, 2010; nccn.org). Participants will rate their present level of distress (on a 0-10 scale, with 0 being no distress, to 10 being the most distressed) and then identify particular stressors in the area of practical problems, family problems, emotional problems, spiritual/religious concerns, physical problems, and any additional stressor as identified by the participant.
Change in Depression level | 10 weeks
  Anxiety and depression are two psychological outcomes commonly reported in caregiving research. The Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983) will be used to measure both concepts reflective of psychological wellbeing in patients and caregivers. The HADS is a reliable and valid instrument, with strong internal consistency for cancer populations. It has been used for patients who are hospitalized or ambulatory patients and for caregivers. It consists of 14 items which are scored on a four-point Likert scale (0-3). Items are recoded and summarized into subscales of anxiety and depression (range 0-21). Participants scoring 11 or higher are considered anxious or depressed.
Caregiver Response to the Caregiving Experience | 10 weeks
  The reaction is either positive (caregiver benefit) or negative (caregiver burden). The caregiver reaction will be assessed using the Caregiver Reaction Assessment (CRA). This 24-item instrument will be used to measure the burden of informal caregiving using a 5-point Likert scale. The CRA consists of five subscales that represent positive and negative burden aspects of caregiving. They include 1) impact on schedule; 2) caregiver's esteem; 3) lack of family support; 4) impact on health; and 5) impact on finances. Positive items are reversed scored. Higher scores indicate greater levels of perceived burden.
Caregiver Mastery | 10 weeks
  The Pearlin & Schooler Mastery Instrument (1978) will be used to assess caregiver mastery. Caregiver mastery refers to the caregivers' perceptions of their ability to meet the challenges of caregiving, to feel in control of the situation, and to use effective problem solving skills. The Pearlin & Schooler Master Instrument is a seven item, five-point Likert scale instrument with a Crohnbach's alpha = 0.73. Scoring is done by summing item scores for a total score (possible range 7-35) with higher scores indicating higher levels of mastery. Examples of items include, "I have little control over the things that happen to me", and "There is little I can do to change many of the important things in my life".

CONTACTS AND LOCATIONS:
Overall Officials: Polly Mazanec, PhD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States